CLINICAL TRIAL: NCT04568837
Title: Postoperative Steroids and Recovery After Spine Fusion
Brief Title: Steroids After Spine Fusion Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jung Yoo, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021169
Record Dates: First submitted 2020-09-21; First posted 2020-09-29 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Spine Fusion
MeSH Terms: interventions — Prednisone; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of two groups: treatment group vs control (no treatment) group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Corticosteroid (Experimental): Participants in this group will receive a daily dose of corticosteroids on postoperative day one and two after spine fusion surgery
  Interventions: Drug: Prednisone 20 Mg
- Control (No Intervention): Participants in this group will receive no steroids on postoperative day one and two after spine fusion surgery.

INTERVENTIONS:
Drug: Prednisone 20 Mg — 20 mg of Prednisone or 1 mL of 4 mg/mL Dexamethasone Sodium Phosphate will be administered each day for participants in the intervention group
  Other Names: Dexamethasone Sodium Phosphate 1 mL 4 mg/mL
  Arms: Corticosteroid

SUMMARY:
This trial studies how well low-dose postoperative corticosteroids (FDA approved) affect patient outcomes (patient reported outcomes, pain medication use, length of stay, major complications, and time to first bowel movement) after thoracic and/or lumbar spine fusion surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES This study aims to compare patient outcomes (patient reported outcomes, pain medication use, length of stay, major complications, and time to first bowel movement) between subjects that receive either 20 mg of PO prednisone or 1 mL of 4 mg/mL of IV dexamethasone sodium phosphate and a control group.

OUTLINE Participants are patients who elect to participate in the study prior to scheduled thoracic and/or lumbar spine fusion surgery at Oregon Health and Science University. Participants undergo their scheduled spine fusion surgery. After surgery, participants are randomized into either the study drug group or the control (non-treatment) group. If randomized into the study drug group, participants will orally take a daily dose of 20 mg of prednisone (1 mL of 4 mg/mL dexamethasone sodium phosphate if unable to tolerate oral administration) on postoperative days one and two.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 50 undergoing thoracic and/or lumbar fusion with a Spine Center surgeon will be included

Exclusion Criteria:

* Patient is already taking chronic steroids
* Patient is pregnant
* Patient is decisionally impaired
* Patient is a prisoner

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-10-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
Morphine equivalent pain medication use over the length of hospitalization | From postoperative admission to discharge, up to 4 weeks
  This will be measured by converting the dosage of the pain medication administered to its equivalent dosage of morphine.
Length of hospital stay after surgery | From postoperative admission to discharge, up to 4 weeks
  This will be measured by taking the total minutes the patient stays in the hospital after surgery from time of admission to time of discharge.
Time to first bowel movement in hospital after surgery | From postoperative admission to discharge, up to 4 weeks
  This will be measured in the total number of minutes from admission after surgery that it takes for the patient to have their first bowel movement recorded.
Number of major complications reported during hospital stay after surgery | From postoperative admission to discharge, up to 4 weeks
  This will be measured in the total number of major complications (any) that occur during the hospital stay after surgery. These include, infection, neurological deficit, myocardial infarction, stroke, pneumonia, pulmonary embolism, and bleeding.
Morphine equivalent pain medication use over the first 48 hours of hospitalization | From postoperative admission to 48 hours after
  This will be measured by converting the dosage of the pain medication administered to its equivalent dosage of morphine.

CONTACTS AND LOCATIONS:
Overall Officials: Jung U Yoo, MD, Principal Investigator — Department of Orthopaedics and Rehabilitation
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No